CLINICAL TRIAL: NCT00924352
Title: Phase I/II Trial of Dasatinib Plus Ixabepilone in 2nd or 3rd Line Metastatic Breast Cancer
Brief Title: Trial of Dasatinib Plus Ixabepilone in 2nd or 3rd Line Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSSMBC0804
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixabepilone + Dasatinib (Experimental): Ixabepilone, for injection 15 mg supplied with diluent for ixabepilone, 8 mL. Dose Level 2;20 mg/m2,Dose Level 1;20 mg/m2,Dose Level 0 (Starting Dose);16 mg/m2,Dose Level - 1;12 mg/m2,Dose Level - 2;12 mg/m2.
  Dasatinib tablets will be administered continuously starting on Day 1, Cycle 1 once daily (QD).Dose Level 2;140 mg QD,Dose Level 1;100 mg QD,Dose Level 0 (Starting Dose);100 mg QD,Dose Level - 1;100 mg QD,Dose Level - 2;70 mg QD.
  Interventions: Drug: Dasatinib; Drug: Ixabepilone

INTERVENTIONS:
Drug: Dasatinib — Dasatinib tablets will be administered continuously starting on Day 1, Cycle 1 once daily (QD).Dose Level 2;140 mg QD,Dose Level 1;100 mg QD,Dose Level 0 (Starting Dose);100 mg QD,Dose Level - 1;100 mg QD,Dose Level - 2;70 mg QD.
  Other Names: SPRYCEL
Drug: Ixabepilone — Ixabepilone, for injection 15 mg supplied with diluent for ixabepilone, 8 mL. Dose Level 2;20 mg/m2,Dose Level 1;20 mg/m2,Dose Level 0 (Starting Dose);16 mg/m2,Dose Level - 1;12 mg/m2,Dose Level - 2;12 mg/m2.
  Other Names: IXEMPRA

SUMMARY:
The primary objective for the Phase I portion of the study is to determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) and for the Phase II portion of the study is to evaluate progression free survival (PFS). Secondary objectives are response rate, clinical benefit rate, and overall toxicity.

DETAILED DESCRIPTION:
In the Phase I portion of the study, patients will receive study treatment according to the assigned dose level. Ixabepilone will be administered over 1 hour on Days 1, 8, and 15 of a 28-day cycle. Dasatinib will be administered continuously starting on Day 1, Cycle 1 once daily (QD).

Three patients will be enrolled at dose level 0 and observed for dose-limiting toxicity (DLT) for 1 course of treatment.

Dose escalation or reduction will depend on the number of patients experiencing DLT as follows:

* If 0 of 3 patients experiences a DLT, then 3 additional patients will be enrolled at the next higher dose level.
* If 1 of 3 patients experiences a DLT, then 3 additional patients will be enrolled at that dose level.
* If 2 of 3 or 3 of 3 patients experience a DLT, then 3 patients will be enrolled at the next lower dose unless 6 patients have already been treated at that dose.
* If ≥2 of 6 patients experience a DLT at that dose level, then the MTD is considered to have been exceeded. At that point, 3 patients are treated at the next lower dose.
* If no more than 1 of the 6 patients experiences a DLT, then the dose level will be escalated 1 level.

Maximum-tolerated dose (MTD) is defined as the dose at which ≤1 of 6 patients experience DLT, and above which ≥2 of 6 patients experience DLT.

In the Phase II portion of the study, dasatinib and ixabepilone will be administered at the MTD determined during Phase I. Dasatinib will be started on Day 1, Cycle 1 and will be administered continuously once daily. Ixabepilone will be administered over 1 hour on Days 1, 8, and 15 of a 28-day cycle. Patients will be treated with both agents for up to 8 cycles, after which stable or responding patients are eligible for monotherapy with dasatinib at the investigator's discretion in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet each of the following criteria to be considered eligible for inclusion in this study:

1. Patient has the ability to understand and the willingness to sign a written informed consent including form according to institutional guidelines.
2. Patient has histologically-proven breast cancer.
3. Patient has locally recurrent or metastatic disease, measurable or non- measurable by RECIST criteria.
4. Patient has HER2-negative disease or disease that is refractory to HER2- directed therapy.
5. Patient is female or male ≥ 18 years of age.
6. Patient has(ECOG)performance status of ≤ 2.
7. Patient must have received at least 1 but no more than 2 prior chemotherapy regimens for locally recurrent or metastatic disease. Patients may have received neoadjuvant and/or adjuvant chemotherapy. These prior regimens can not have included ixabepilone or dasatinib. A line of chemotherapy will be defined as one or more agents used continuously or discontinuously (i.e., allowing a break or chemo holiday) without the addition of a new agent. Hormonal therapy will not be considered a line of therapy.
8. Prior chemotherapy must have been completed at least 3 weeks prior to study treatment start (6 weeks for nitrosoureas and mitomycin), and the patient must have recovered from all associated toxicities (except for alopecia and neuropathy grade 1 according to CTCAE, v3.0 classification).
9. Radiation therapy, immunotherapy, biologic therapy, and hormonal/endocrine therapy must have been completed at least 2 weeks prior to study treatment start. Any major surgery must have been completed at least 4 weeks prior to study treatment start.
10. Patient has adequate organ, metabolic and bone marrow function as follows:

    1. Total bilirubin ≤ 1.0 × institutional ULN
    2. AST, ALT ≤ 2.5 × institutional ULN
    3. Serum sodium, potassium, calcium, magnesium, and phosphate ≥ institutional LLN. (Hypokalemia or hypomagnesemia must be corrected prior to dasatinib administration.)
    4. Serum creatinine < 1.5 × institutional ULN
    5. Hematologic function: - ANC ≥ 1500/mm3. -Platelet count ≥ 100,000/mm3. - Hemoglobin ≥ 10.0 g/dL
    6. PT and PTT < 1.5 x institutional ULN
11. Ability to take oral medication (dasatinib must be swallowed whole).
12. Concomitant medications:

    1. Patient agrees to discontinue St John's Wort at least 5 days prior to starting dasatinib therapy and while receiving dasatinib therapy.
    2. Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
    3. The use of CYP3A4 inducers, inhibitors, and substrates; medications that prolong QT interval; antacids; H2 blockers and proton pump inhibitors; and medications that inhibit platelet function and anticoagulation should be avoided during dasatinib therapy. These are restricted therapies that are permitted with caution when medically indicated.
13. Women of childbearing potential must have a negative serum or urine pregnancy test prior to the start of study treatment.
14. Patients of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study treatment is stopped.

Exclusion Criteria:

A patient who meets any of the following criteria will be considered not eligible for inclusion in this study:

1. Patient has had prior treatment with ixabepilone, dasatinib, or both.
2. Patient has had more than 2 prior lines of chemotherapy for locally recurrent or metastatic breast cancer. A line of chemotherapy will be defined as one or more agents used continuously or discontinuously (i.e., allowing a break or chemo holiday) without the addition of a new agent. Hormonal therapy will not be considered a line of therapy.
3. Patient has received a cumulative dose of > 360 mg/m2 of doxorubicin or > 600 mg/m2 of epirubicin.
4. Prior radiation must not have included ≥ 30% of major bone marrow containing areas (pelvis, lumbar spine).
5. Patients with CTC grade 2 or greater neuropathy (motor or sensory) at study entry.
6. Patient has evidence CNS or brain metastases, unless CNS or brain metastases have been treated and stable for > 3 months.
7. Patient has psychiatric illness or social situation that would limit or prohibit compliance with study requirements.
8. Patient has an inability to take oral medication or inability to absorb oral medication.
9. Patient has had any invasive cancer other than the one being treated in this study within 3 years with the exception of surgically cured nonmelanoma skin cancer; in situ carcinoma of the cervix; in situ carcinoma of the breast.
10. Patient is receiving concurrent cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, or hormonal therapy for cancer).
11. Patient has other serious medical conditions as judged by the Principal Investigator.
12. Patient has a concurrent medical condition which may increase the risk of toxicity.
13. Patient has a pleural or pericardial effusion of any grade.
14. Patient has cardiac symptoms including any of the following:

    1. Uncontrolled angina, congestive heart failure or myocardial infarction within 6 months of study entry.
    2. Diagnosed congenital long QT syndrome.
    3. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).
    4. Prolonged QTc on pre-entry ECG (> 450 msec).
    5. Hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration.
15. Patient has a history of significant bleeding disorder unrelated to cancer, including:

    1. Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease).
    2. Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).
    3. Ongoing or recent (≤ 3 months) significant GI bleeding.
16. Patient is taking any of the following concomitant medications at study entry:

    a. Category I drugs that are generally accepted to have a risk of causing Torsades de pointes including (Patients must discontinue drug 7 days prior to starting dasatinib.):
    * quinidine, procainamide, disopyramide.
    * amiodarone, sotalol, ibutilide, dofetilide.
    * erythromycin, clarithromycin.
    * chlorpromazine,haloperidol,mesoridazine, thioridazine,pimozide .
    * cisapride,bepridil, droperidol, methadone, arsenic, chloroquine, domperidone,halofantrine, levomethadyl, pentamidine,sparfloxacin, lidoflazine.
17. Patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ixabepilone or dasatinib. Ixabepilone is contraindicated in patients who have a known, prior, severe (CTC grade 3 or 4) history of hypersensitivity reaction to a drug formulated in Cremophor® EL (polyoxyethylated castor oil).
18. Patient has received any investigational agent or therapy within 30 days prior to study treatment start.
19. Patient is unwilling or unable to comply with study requirements.
20. Women who:

    1. are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study treatment, or
    2. have a positive pregnancy test at baseline, or
    3. are pregnant or breastfeeding.
21. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Schwartzberg, MD, FACP, Study Chair — The West Clinic
Locations (13):
- United States (13):
  - Hematology Oncology PC, Stamford, Connecticut
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - North Shore Cancer Research, Skokie, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Baystate Medical Center, Springfield, Massachusetts
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Oncology Hematology Specialists, P.A., Denville, New Jersey
  - The Moses H. Cone Regional Cancer Center, Greensboro, North Carolina
  - North Coast Cancer Care, Sandusky, Ohio
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Phase I portion of this study was conducted at 4 oncology clinics located in the United States. The Phase II portion of the study was conducted at the 4 Phase I sites, plus 10 additional oncology clinics located in the United States. Enrollment started in July 2009 and was completed in June 2012.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent screening procedures to verify eligibility.
Groups:
- Phase I: The Phase I sample includes patients who were enrolled into the Phase I portion of this study. Patients received treatment according to the assigned dose level. Ixabepilone was administered over 1 hour on Days 1, 8, and 15 of a 28-day cycle. Dasatinib was administered continuously starting on Day 1, Cycle 1 once daily. Patients were treated with both agents for up to 8 cycles, after which stable or responding patients were eligible for dasatinib monotherapy at the investigator's discretion in the absence of disease progression or unacceptable toxicity.
- Phase II: The Phase II sample includes patients who were enrolled into the Phase II portion of this study. Dasatinib and ixabepilone were administered at the maximum tolerated dose determined during the Phase I portion: dasatinib 100 mg daily and ixabepilone 20 mg/m2. Ixabepilone was administered over 1 hour on Days 1, 8, and 15 of a 28-day cycle. Dasatinib was administered continuously starting on Day 1, Cycle 1 once daily. Patients were treated with both agents for up to 8 cycles, after which stable or responding patients were eligible for dasatinib monotherapy at the investigator's discretion in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 12 | 44
Completed | 12 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone + Dasatinib: Ixabepilone, for injection 15 mg supplied with diluent for ixabepilone, 8 mL. Dose Level 2;20 mg/m2,Dose Level 1;20 mg/m2,Dose Level 0 (Starting Dose);16 mg/m2,Dose Level - 1;12 mg/m2,Dose Level - 2;12 mg/m2.
  Dasatinib tablets will be administered continuously starting on Day 1, Cycle 1 once daily (QD).Dose Level 2;140 mg QD,Dose Level 1;100 mg QD,Dose Level 0 (Starting Dose);100 mg QD,Dose Level - 1;100 mg QD,Dose Level - 2;70 mg QD.
  Dasatinib: Dasatinib tablets will be administered continuously starting on Day 1, Cycle 1 once daily (QD).Dose Level 2;140 mg QD,Dose Level 1;100 mg QD,Dose Level 0 (Starting Dose);100 mg QD,Dose Level - 1;100 mg QD,Dose Level - 2;70 mg QD.
  Ixabepilone: Ixabepilone, for injection 15 mg supplied with diluent for ixabepilone, 8 mL.
  Dose Level 2;20 mg/m2,Dose Level 1;20 mg/m2,Dose Level 0 (Starting Dose);16 mg/m2,Dose Level - 1;12 mg/m2,Dose Level - 2;12 mg/m2.
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) of Dasatinib When Given in Combination With Ixabepilone (Phase I)
Description: The MTD of dasatinib (taken daily, continuously) when given in combination with ixabepilone (administered on Days 1, 8, and 15 of a 28-day cycle) was determined using a standard 3 + 3 dose escalation cohort design. The total sample and the number of patients who receive each dose in this design depends on the frequency of dose limiting toxicities (DLT) at each dosage. The MTD was defined as the dose at which ≤ 1 of 6 patients experienced DLT, and above which ≥ 2 of 6 patients experienced DLT.
Time Frame: MTD was assessed during the first cycle of combination therapy (days 1-28).
Population: The Phase I analysis sample includes the 12 patients who were enrolled into the Phase I portion of the study.
Measure: Number; unit: mg daily
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 12
mg daily | 100

2. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) of Ixabepilone When Given in Combination With Dasatinib (Phase I)
Description: The MTD of ixabepilone (administered on Days 1, 8, and 15 of a 28-day cycle) when given in combination with dasatinib (taken daily, continuously) was determined using a standard 3 + 3 dose escalation cohort design. The total sample and the number of patients who receive each dose in this design depends on the frequency of dose limiting toxicities (DLT) at each dosage. The MTD was defined as the dose at which ≤ 1 of 6 patients experienced DLT, and above which ≥ 2 of 6 patients experienced DLT.
Time Frame: MTD was assessed during the first cycle of combination therapy (days 1-28).
Population: The Phase I analysis sample includes the 12 patients who were enrolled into the Phase I portion of the study.
Measure: Number; unit: mg/m2
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 12
mg/m2 | 20

3. Primary Outcome: Determination of the Dose Limiting Toxicities (DLTs) of the Combination of Dasatinib and Ixabepilone (Phase I)
Description: DLTs were assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Dose limiting toxicity was defined as any grade 4 hematologic event or any grade 3 or 4 non-hematologic event occurring during cycle 1 that is attributable to dasatinib, ixabepilone, or the combination. The following events were excluded from this definition: grade 4 neutropenia lasting for 3 days or less; grade 3 nausea responsive to antiemetics; grade 3 infection with normal ANC or grade 1 or 2 neutrophils; grade 3 diarrhea responsive to optimal use of antidiarrheal therapy.
Time Frame: DLTs were assessed during the first cycle of combination therapy (days 1-28).
Population: The Phase I analysis sample includes the 12 patients who were enrolled into the Phase I portion of the study.
Measure: Number; unit: participants
Groups:
- Ixabepilone + Dasatinib (Dose Level 0): Dasatinib 100 mg daily and Ixabepilone 16 mg/m2 on Days 1, 8, and 15 of a 28-day cycle.
- Ixabepilone + Dasatinib (Dose Level 1): Dasatinib 100 mg daily and Ixabepilone 20 mg/m2 on Days 1, 8, and 15 of a 28-day cycle.
- Ixabepilone + Dasatinib (Dose Level 2): Dasatinib 140 mg daily and Ixabepilone 20 mg/m2 on Days 1, 8, and 15 of a 28-day cycle.
Arm/Group | Ixabepilone + Dasatinib (Dose Level 0) | Ixabepilone + Dasatinib (Dose Level 1) | Ixabepilone + Dasatinib (Dose Level 2)
Number analyzed (Participants) | 3 | 6 | 3
participants
  DLT: Grade 4 Thrombocytopenia | 0 | 0 | 1
  DLT: Grade 4 Leukopenia | 0 | 0 | 1

4. Secondary Outcome: Best Overall Response of the Combination of Dasatinib and Ixabepilone (Phase II)
Description: Best overall response is defined as the best response across all time points. Response was evaluated via changes from baseline in radiological tumor measurements performed after every two treatment cycles and at the end of treatment or time of progression. Response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: Response to treatment was assessed after about every 8 weeks of treatment, for up to 27.2 months.
Population: The Phase II analysis sample of 50 patients includes the 6 patients from the Phase I portion of the study who were treated at the MTD as well as the 44 patients who were enrolled into the Phase II portion of the study.
Measure: Number; unit: participants
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 50
participants
  Complete Response | 0
  Partial Response | 4
  Stable Disease | 11
  Progressive Disease | 23
  Not Evaluable | 12

5. Secondary Outcome: Clinical Benefit Rate of the Combination of Dasatinib and Ixabepilone (Phase II)
Description: Clinical benefit rate was defined as the percentage of participants experiencing stable disease (SD) of at least 24 weeks (from the start of treatment) plus complete response (CR) and partial response (PR). Response was evaluated via changes from baseline in radiological tumor measurements performed after every two treatment cycles and at the end of treatment or time of progression. Response was evaluated using RECIST version 1.0 guidelines, where CR is the disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter(LD) of target lesions; SD is neither sufficient shrinkage in sum of longest diameter of target lesions to be PR nor increase of >=20%.
Time Frame: Response to treatment was assessed after about every 8 weeks of treatment, for up to 27.2 months.
Measure: Number; unit: percentage of participants
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 50
percentage of participants | 26.0

6. Secondary Outcome: Incidence of Grade 3 Adverse Events (AEs) With the Combination of Dasatinib and Ixabepilone (Phase II)
Description: All treatment emergent adverse events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: Adverse events were collected beginning on day 1 of treatment until one month after the end of study treatment.
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 50
participants | 31

7. Secondary Outcome: Incidence of Grade 4 Adverse Events (AEs) With the Combination of Dasatinib and Ixabepilone (Phase II)
Description: as for outcome 6
Time Frame: Adverse events were collected beginning on day 1 of treatment until one month after the end of study treatment.
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 50
participants | 5

8. Primary Outcome: Evaluation of Progression-free Survival (PFS) of the Combination of Dasatinib and Ixabepilone (Phase II)
Description: Disease progression was determined through radiology imaging measurements and by clinical or symptomatic progression during or after treatment. Progression is defined per RECIST v1.0 guidelines as a measurable increase in the smallest diameter of any target lesion, progression of existing non-target lesions, or the appearance of 1 or more new lesions.
Time Frame: PFS was measured from day 1 of treatment until time of progression (assessed about every 8 weeks) or death, whichever came first, for up to 27.2 months.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone + Dasatinib
Number analyzed (Participants) | 50
months | 6.01 [2.92 to 8.08]

ADVERSE EVENTS:
Time Frame: Adverse events were collected on day 1 of treatment until one month after the end of study treatment.
Arm/Group | Ixabepilone + Dasatinib
Serious Adverse Events (participants affected / at risk) | 11/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone + Dasatinib (N=56)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Edema due to Cardiac Disease (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Electrocardiogram QT Prolonged (Investigations) | 1
QT Prolonged (Investigations) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone + Dasatinib (N=56)
Anemia (Blood and lymphatic system disorders) | 29
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 8
White Blood Cell Disorder (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 3
Sinus Tachycardia (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Eye Irritation (Eye disorders) | 1
Eyelid Edema (Eye disorders) | 1
Vision Blurred (Eye disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 7
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 31
Dry Mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 30
Salivary Hypersecretion (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 22
Asthenia (General disorders) | 3
Chest Pain (General disorders) | 2
Chills (General disorders) | 3
Fatigue (General disorders) | 34
Generalized Edema (General disorders) | 1
Influenza-like Illness (General disorders) | 1
Infusion-related Reaction (General disorders) | 1
Injection Site Pain (General disorders) | 1
Localized Edema (General disorders) | 1
Malaise (General disorders) | 1
Mucosal Inflammation (General disorders) | 1
Mucosal Ulceration (General disorders) | 1
Myalgia (General disorders) | 1
Nodule (General disorders) | 1
Edema (General disorders) | 1
Edema Peripheral (General disorders) | 4
Pain (General disorders) | 2
Pyrexia (General disorders) | 8
Hyperbilirubinemia (Hepatobiliary disorders) | 1
Cytokine Release Syndrome (Immune system disorders) | 2
Hypersensitivity (Immune system disorders) | 3
Breast Infection (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Eye Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tooth Abscess (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 5
Vulvovaginal Mycotic Infection (Infections and infestations) | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Infusion-related Reaction (Injury, poisoning and procedural complications) | 4
Muscle Strain (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Wound Complication (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 5
Blood Alkaline Phosphatase Increased (Investigations) | 2
Blood Creatinine Increased (Investigations) | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1
Electrocardiogram QT Prolonged (Investigations) | 2
Hemoglobin Decreased (Investigations) | 6
Neutrophil Count (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 3
Platelet Count Decreased (Investigations) | 1
QT Prolonged (Investigations) | 2
Weight Decreased (Investigations) | 4
White Blood Cell Count (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 3
Decreased Appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1
Ocular Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 18
Headache (Nervous system disorders) | 17
Hypoesthesia (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 20
Paresthesia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Photophobia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 7
Confusional State (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 7
Mood Altered (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Micturition Urgency (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Breast Pain (Reproductive system and breast disorders) | 1
Nipple Pain (Reproductive system and breast disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 12
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1
Hair Disorder (Skin and subcutaneous tissue disorders) | 1
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 12
Rash Generalized (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 2
Skin Disorder (Skin and subcutaneous tissue disorders) | 1
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 2
Swelling Face (Skin and subcutaneous tissue disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Epistaxis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The funder will be provided with a copy of the proposed publication at least 30 days prior to its submission or presentation. The funder may request the presentation/submission be delayed for an additional 90 days to allow the funder to seek patent protection. The funder can require the deletion of information deemed as confidential.